CLINICAL TRIAL: NCT04112849
Title: Electronic S3 Prediction of Hospital Readmissions for Heart Failure Exacerbation
Brief Title: Electronic S3 Prediction of Hospital Readmissions for HF Exacerbation
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY12419
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Heart failure subjects: Subjects who have heart failure, and meet inclusion/exclusion criteria, who will be enrolled in this study and will have their heart sounds measured with Nanowear vest (NCHFMS).
  Interventions: Diagnostic Test: Measurement of S3 heart sound

INTERVENTIONS:
Diagnostic Test: Measurement of S3 heart sound — S3 heart sound to be measured by Nanowear Congestive Heart Failure Management System device.

SUMMARY:
The study objective is to measure the value of the third heart sound (S3) for the prediction of recurrent heart failure (HF). For the purpose of this study, a heart failure event will be defined as a hospitalization with a primary diagnosis of heart failure. The main hypothesis of the study is that measurement of S3, using a microelectronic machine microphone positioned in a wearable device (Nanowear Wearable Congestive Heart Failure Management System) near the time of discharge from a hospitalization for heart failure, can predict which patients will be at high risk for a heart failure event, thereby identifying a group in whom increased surveillance and monitoring may decrease hospital readmissions for worsening heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is a complex clinical syndrome that results from any structural or functional impairment of the heart that affects the filling or ejection of blood in a cardiac cycle. HF manifests clinically as fatigue and dyspnea (shortness of breath). This may in turn result in exercise intolerance and fluid retention. Fluid retention leads to pulmonary congestion and/or peripheral edema [Yancy, 2017]. Cardiac rhythm abnormalities are very common among HF patients. Any new abnormalities that arise in a patient with fluid decompensation prolongs hospitalization as well as increases mortality rates [Lloyd-Jones, 2010; Ross, 2009; Chaudhry, 2015].

Within 5 years of a HF diagnosis, the mortality rate is 50%. The 30 day, 1-year and 5-year mortality rates after HF related hospitalization were 10.4%, 22 % and 42.3 % respectively. Post discharge mortality increased from 4.3% to 6.4% between 1993 and 2005 [Lloyd-Jones, 2010; Ross, 2009]. In 2006, the number of deaths with a mention of HF was as high as it was in 1995. 1 out of every 9 mortalities in the US has HF mentioned as a cause. HF related deaths are approximately 7% of all cardiovascular diseases. In the US, HF related costs exceeded $30 billion in 2013. The average cost per patient for HF related hospitalization was $23,077. Hospitalization after a HF diagnosis happens at least once in 83% of the patients and up to four times in 43% of the patients [Yancy, 2017; Lloyd-Jones, 2010; Ross, 2009].

Heart sounds, and particularly the third heart sound, are well known as specific a very specific clinical signs for heart failure and are associated with worse clinical outcomes. In the context of HF the presence of a pronounced or audible S3 is a specific sign of elevated filling pressures and is suggestive of a restrictive filling pattern with a steep transmitral E-wave [Siejko, 2017]. Recent advances in digital audio technology allow us to not simply assess for the presence or absence of a third heart in objective measures, but also allow us to quantitate it [Buck, 2017; Adamson, 2014; Lloyd, 2019]. Further, recent work has demonstrated that if a frequency range to detect and quantitate the third heart sound is used that extends below the usual range for human hearing, that the third heart sound may be even more predictive of clinical outcomes. The investigators are working with a device manufacturer who have a wearable diagnostic device that includes a directional microelectronic machine microphone that can effectively detect heart sounds. This device will be used to detect and quantitate heart sounds, and specifically the third heart sound, to investigate the prognostic implications of a third heart sound.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion 1. Subject has provided informed consent
* Inclusion 2. Male or female over the age of 18 years
* Inclusion 3. The patient is either hospitalized with a primary diagnosis of acute heart failure or was discharged with a primary diagnosis of acute heart failure within 2 weeks prior to enrollment.
* Inclusion 4. NYHA functional class II-IV at time of enrollment
* Inclusion 5. Subjects were patients of Penn State Hershey Medical Center (PSHMC), who are/were admitted at PSHMC.

Exclusion Criteria:

* Exclusion 1. Subject unwilling or unable to wear the system for one measurement prior to discharge or within the first two weeks following discharge.
* Exclusion 2. Subjects who are limited by angina.
* Exclusion 3. Severe aortic stenosis.
* Exclusion 4. Subjects who are hemodynamically unstable requiring support with intravenous vasoactive medications or mechanical circulatory support
* Exclusion 5. Symptomatic ventricular arrhythmias within the past 6 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, 18 and older, admitted to the hospital with a primary diagnosis of acute heart failure and NYHA class II-IV at time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of hospital readmissions for heart failure | 90 days from initial hospitalization for acute heart failure
  Total hospitalizations will be monitored from time patient is initially discharged for acute heart failure until 90 days post-discharge.

SECONDARY OUTCOMES:
New York Heart Association (NYHA) functional class during hospital readmissions for heart failure | 90 days from initial hospitalization for acute heart failure
  If applicable, New York Heart Association (NYHA) functional class will be assessed during readmission for heart failure. NYHA Functional Classification places patients in one of four categories based on how much they are limited during physical activity; Class I being best and Class IV being the worst functional class. Class I has no limitation to physical activity, Class II has slight limitation to physical activity, Class III has marked limitation of physical activity, and Class IV is unable to carry out any physical activity without severe discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: John Boehmer, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Card Fail. 2017 Aug;23(8):628-651. doi: 10.1016/j.cardfail.2017.04.014. Epub 2017 Apr 28. No abstract available. PMID 28461259
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Ross JS, Chen J, Lin Z, Bueno H, Curtis JP, Keenan PS, Normand SL, Schreiner G, Spertus JA, Vidan MT, Wang Y, Wang Y, Krumholz HM. Recent national trends in readmission rates after heart failure hospitalization. Circ Heart Fail. 2010 Jan;3(1):97-103. doi: 10.1161/CIRCHEARTFAILURE.109.885210. Epub 2009 Nov 10. PMID 19903931
- [Background] Chaudhry SI, Wang Y, Concato J, Gill TM, Krumholz HM. Patterns of weight change preceding hospitalization for heart failure. Circulation. 2007 Oct 2;116(14):1549-54. doi: 10.1161/CIRCULATIONAHA.107.690768. Epub 2007 Sep 10. PMID 17846286
- [Background] Siejko KZ, Thakur PH, Maile K, Patangay A, Olivari MT. Feasibility of heart sounds measurements from an accelerometer within an ICD pulse generator. Pacing Clin Electrophysiol. 2013 Mar;36(3):334-46. doi: 10.1111/pace.12059. Epub 2012 Dec 17. PMID 23252962
- [Background] Lloyd T, Buck H, Foy A, Black S, Pinter A, Pogash R, Eismann B, Balaban E, Chan J, Kunselman A, Smyth J, Boehmer J. The Penn State Heart Assistant: A pilot study of a web-based intervention to improve self-care of heart failure patients. Health Informatics J. 2019 Jun;25(2):292-303. doi: 10.1177/1460458217704247. Epub 2017 May 14. PMID 28504048
- [Background] Buck H, Pinter A, Poole E, Boehmer J, Foy A, Black S, Lloyd T. Evaluating the older adult experience of a web-based, tablet-delivered heart failure self-care program using gerontechnology principles. Geriatr Nurs. 2017 Nov-Dec;38(6):537-541. doi: 10.1016/j.gerinurse.2017.04.001. Epub 2017 May 26. PMID 28554497
- [Background] Adamson PB, Smith AL, Abraham WT, Kleckner KJ, Stadler RW, Shih A, Rhodes MM; InSync III Model 8042 and Attain OTW Lead Model 4193 Clinical Trial Investigators. Continuous autonomic assessment in patients with symptomatic heart failure: prognostic value of heart rate variability measured by an implanted cardiac resynchronization device. Circulation. 2004 Oct 19;110(16):2389-94. doi: 10.1161/01.CIR.0000139841.42454.78. Epub 2004 Aug 16. PMID 15313946